CLINICAL TRIAL: NCT03251664
Title: The Relation of Locally Available Food Items With Anemia Status Among Pregnant Women in Ethiopia
Brief Title: Food Groups Associated With Anaemia in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shimels Hussien Mohammed, Community Nutrition Researcher, Tehran University of Medical Sciences
Other Study IDs: AAHB-217/15
Record Dates: First submitted 2017-08-12; First posted 2017-08-16 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Anemia; Dietary Habits; Food Habits
MeSH Terms: conditions — Anemia; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anemic: Hemoglobin <11 g/l
  Interventions: Dietary Supplement: Food groups consumed
- Non-anemic: Hemoglobin 11 g/l (and above)
  Interventions: Dietary Supplement: Food groups consumed

INTERVENTIONS:
Dietary Supplement: Food groups consumed

SUMMARY:
This study investigates the association between locally consumed food items with anemia among pregnant women, in Addis Ababa city, Ethiopia.

DETAILED DESCRIPTION:
Prevention of anemia among women, particularly pregnant women, is a priority nutrition agenda in Ethiopia. Anemia is a significant contributor to poor pregnancy outcomes, including low birth weight and maternal mortality. Anemia is of multiple influences, which in most of the cases include dietary factors. Consumption food items rich in iron and other nutrients involved in red blood cell production promotes optimal hemoglobin level. Dark green leafy vegetables, meat, and beans are some of the food groups reported to be associated with lesser risk of anemia. Studies on the relation of indigenous food items with health outcome are limited in developing countries. For example, teff, consumed only in Ethiopia and parts of Eritrea, is traditionally believed to be protective of anemia because of its high iron content, but Khat chewing, a pervasive social practice in Ethiopia, has been associated with restrictive eating pattern and anemia. In this study, the association of locally consumed food groups with anemia was investigated among pregnant Ethiopian women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Age 18 years and above
* Residence in Addis Ababa city

Exclusion Criteria:

* Serious medical illness

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women in Addis Ababa city, Ethiopia
Sampling Method: Probability Sample
Enrollment: 592 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-02-20 (Actual); Study Completion 2016-02-20 (Actual)

PRIMARY OUTCOMES:
Food items/groups association with anemia | October 2015 to February 2016
  Relation of food groups with anemia risk

SECONDARY OUTCOMES:
Reproductive factors associated with anemia | October 2015 to February 2016
  Relation of reproductive and obstetrics history with anemia
Sociodemographic and economic factors association with anemia | October 2015 to February 2016
  Relation of socioeconomic factors with anemia

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Esmaillzadeh, PhD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Addis Ababa Health Bureau, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided.

REFERENCES:
- [Derived] Mohammed SH, Taye H, Larijani B, Esmaillzadeh A. Food taboo among pregnant Ethiopian women: magnitude, drivers, and association with anemia. Nutr J. 2019 Mar 23;18(1):19. doi: 10.1186/s12937-019-0444-4. PMID 30904017
- [Derived] Mohammed SH, Taye H, Sissay TA, Larijani B, Esmaillzadeh A. Teff consumption and anemia in pregnant Ethiopian women: a case-control study. Eur J Nutr. 2019 Aug;58(5):2011-2018. doi: 10.1007/s00394-018-1759-1. Epub 2018 Jun 23. PMID 29936535